CLINICAL TRIAL: NCT01784718
Title: Compassionate Use of Buphenyl® in the Treatment of Byler's Disease
Brief Title: Buphenyl Therapy for Byler's Disease
Status: No longer available | Type: Expanded Access
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO12070385
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Byler Disease
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1 | interventions — 4-phenylbutyric acid

INTERVENTIONS:
Drug: Buphenyl

SUMMARY:
This is a single patient compassionate use protocol to determine whether Buphenyl (4-phenylbutyrate) will improve the poor bile flow associated with Byler Disease.

ELIGIBILITY:
Inclusion Criteria:

* Byler Disease
* Cholestasis unresponsive to pharmacologic therapy

Exclusion Criteria:

* Allergy/Hypersensitivity to Buphenyl

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult